CLINICAL TRIAL: NCT03935919
Title: Perioperative Continuous Glucose Monitoring in Patients Undergoing an Abdominal Surgery - an Observational Study
Brief Title: Perioperative Continuous Glucose Monitoring in Patients Undergoing an Abdominal Surgery
Acronym: GluPop
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: GluPop
Record Dates: First submitted 2019-04-28; First posted 2019-05-02 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus; Prediabetes
Keywords: perioperative glucose management; continuous glucose monitoring; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study it to assess whether the continuous glucose monitor system Dexcom G6® can be reliably used for perioperative glucose monitoring in 20 prediabetic or diabetic patients undergoing abdominal surgery in terms of data continuity, accuracy and patient tolerability.

DETAILED DESCRIPTION:
The current recommended method for monitoring glucose control is bedside point of care capillary blood glucose testing. A significant limitation for this method is the frequency by which blood glucose testing is typically performed, at most 4-6 times daily. Continuous glucose monitoring (CGM) provides an alternative approach to measure glucose values with the advantage of greater frequency of monitoring as it is measured every few minutes.

Whilst CGM use in the outpatient setting is rising and has demonstrated benefits on glycaemic control, the accuracy of these devices perioperatively is less investigated. In this study the sixth-generation factory-calibrated real-time Dexcom G6® system will be used as a CGM and its glucose values perioperatively will be compared to the capillary glucose values which will be measured simultaneously by the Accu-Check Inform II (Roche Diagnostics) point-of-care blood glucose meter.

The Investigators aim to assess the feasibility and accuracy of perioperative CGM.

ELIGIBILITY:
Inclusion criteria:

* Aged ≥18 years
* Pre-diabetic (HbA1c 5.7-6.5%) or diabetic (regardless of aetiology)
* Scheduled to have elective abdominal surgery at the University Hospital Bern
* Surgery duration >2 hours

Exclusion criteria:

* Planned MRI procedure during hospitalization
* Inability to follow procedures
* Incapacity to give informed consent
* Presence of extensive skin abnormalities at the sensor insertion site (upper arm)
* Known allergic/irritative skin reactions to dressings/adhesives
* Haematocrit values outside the normal range
* Patients with immunosuppression defined as neutrophil count <0.5x10^9/L
* Patients on isolation precautions (contact, droplet, airborne)
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve a total of 20 adults with pre-diabetes, type 1 or type 2 diabetes who will undergo elective abdominal surgery at the University Hospital Bern.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Sensor accuracy in the perioperative period | 1 day
  Mean Absolute Relative Difference (MARD) between Dexcom G6 sensor glucose values and capillary blood glucose values measured using the Accu-Check Inform II meter in the perioperative period (%)

SECONDARY OUTCOMES:
Mean absolute relative difference between sensor glucose and reference glucose in the preoperative period (%) | 1 week
  Mean absolute relative difference between sensor glucose and reference glucose (for reference values >3.9 and <10.0mmol/l, for reference values ≤3.9mmol/l, for reference values ≥10.0mmol/l) in the preoperative period (%)
Mean absolute relative difference between sensor glucose and reference glucose in the postoperative period (%) | 1-2 weeks
  Mean absolute relative difference between sensor glucose and reference glucose (for reference values >3.9 and <10.0mmol/l, for reference values ≤3.9mmol/l, for reference values ≥10.0mmol/l) in the postoperative period (%)
Median absolute relative difference between sensor glucose and reference glucose in the preoperative period (%) | 1 week
  Median absolute relative difference between sensor glucose and reference glucose (for reference values >3.9 and <10.0mmol/l, for reference values ≤3.9mmol/l, for reference values ≥10.0mmol/l) in the preoperative period (%)
Median absolute relative difference between sensor glucose and reference glucose in the perioperative period (%) | 1 day
  Median absolute relative difference between sensor glucose and reference glucose (for reference values >3.9 and <10.0mmol/l, for reference values ≤3.9mmol/l, for reference values ≥10.0mmol/l) in the perioperative period (%)
Median absolute relative difference between sensor glucose and reference glucose in the postoperative period (%) | 1-2 weeks
  Median absolute relative difference between sensor glucose and reference glucose (for reference values >3.9 and <10.0mmol/l, for reference values ≤3.9mmol/l, for reference values ≥10.0mmol/l) in the postoperative period (%)
Percentage of sensor measurements in the preoperative period within the limits specified by the International Organization of Standardization (ISO) : 15197:2013 criteria | 1 week
  Proportion of sensor measurements in the preoperative period within ±15% of reference glucose if the reference value is ≥5.6mmol/l and within 0.8mmol/l if the reference values is <5.6mmol/l (%)
Percentage of sensor measurements in the perioperative period within the limits specified by the ISO: 15197:2013 criteria | 1 day
  Proportion of sensor measurements in the perioperative period within ±15% of reference glucose if the reference value is ≥5.6mmol/l and within 0.8mmol/l if the reference values is <5.6mmol/l (%)
Percentage of sensor measurements in the postoperative period within the limits specified by the ISO: 15197:2013 criteria | 1-2 weeks
  Proportion of sensor measurements in the postoperative period within ±15% of reference glucose if the reference value is ≥5.6mmol/l and within 0.8mmol/l if the reference values is <5.6mmol/l (%)
Bias and 95% limits of agreement of sensor glucose compared to reference glucose in the preoperative period | 1 week
  Calculation of bias and 95% limits of agreement of sensor glucose compared to reference glucose in the preoperative period
Bias and 95% limits of agreement of sensor glucose compared to reference glucose in the perioperative period | 1 day
  Calculation of bias and 95% limits of agreement of sensor glucose compared to reference glucose in the perioperative period
Bias and 95% limits of agreement of sensor glucose compared to reference glucose in the postoperative period | 1-2 weeks
  Calculation of bias and 95% limits of agreement of sensor glucose compared to reference glucose in the postoperative period
Clarke error grid analysis in the preoperative period | 1 week
  Proportion of sensor glucose values in Clark's error grid zones (A, B, A+B, C, D, E)in the preoperative period (%)
Clarke error grid analysis in the perioperative period | 1 day
  Proportion of sensor glucose values in Clark's error grid zones (A, B, A+B, C, D, E) in the perioperative period (%)
Clarke error grid analysis in the postoperative period | 1-2 weeks
  Proportion of sensor glucose values in Clark's error grid zones (A, B, A+B, C, D, E) in the postoperative period (%)
Sensor availability in the preoperative period (%) | 1 week
  Proportion of study period with available sensor glucose values in the preoperative period
Sensor availability in the perioperative period (%) | 1 day
  Proportion of study period with available sensor glucose values in the perioperative period
Sensor availability in the postoperative period (%) | 1-2 weeks
  Proportion of study period with available sensor glucose values in the postoperative period
Number of sensor replacement events in the preoperative period | 1 week
  Number of times that the sensor needed to be replaced in the preoperative period
Number of sensor replacement events in the perioperative period | 1 day
  Number of times that the sensor needed to be replaced in the perioperative period
Number of sensor replacement events in the postoperative period | 1-2 weeks
  Number of times that the sensor needed to be replaced in the postoperative period
Number of adverse device effects in the preoperative period | 1 week
  Adverse event related to the use of study devices (e.g. skin irritative and allergic reactions, bleeding) in the preoperative period
Number of adverse device effects in the perioperative period | 1 day
  Adverse event related to the use of study devices (e.g. skin irritative and allergic reactions, bleeding) in the perioperative period
Number of adverse device effects in the postoperative period | 1-2 weeks
  Adverse event related to the use of study devices (e.g. skin irritative and allergic reactions, bleeding) in the postoperative period
Percentage of time in the preoperative period with sensor glucose levels within target range | 1 week
  Proportion of time in the preoperative period with sensor glucose levels between 3.9-10.0mmol/l
Percentage of time in the perioperative period with sensor glucose levels within target range | 1 day
  Proportion of time in the perioperative period with sensor glucose levels between 3.9-10.0mmol/l
Percentage of time in the postoperative period with sensor glucose levels within target range | 1-2 weeks
  Proportion of time in the postoperative period with sensor glucose levels between 3.9-10.0mmol/l
Percentage of time in the preoperative period with sensor glucose levels below target range | 1 week
  Proportion of time in the preoperative period with sensor glucose levels below 3.9mmol/l
Percentage of time in the perioperative period with sensor glucose levels below target range | 1 day
  Proportion of time in the perioperative period with sensor glucose levels below 3.9mmol/l
Percentage of time in the postoperative period with sensor glucose levels below target range | 1-2 weeks
  Proportion of time in the postoperative period with sensor glucose levels below 3.9mmol/l
Percentage of time in the preoperative period with sensor glucose levels above target range | 1 week
  Proportion of time in the preoperative period with sensor glucose levels above 10.0mmol/l
Percentage of time in the perioperative period with sensor glucose levels above target range | 1 day
  Proportion of time in the perioperative period with sensor glucose levels above 10.0mmol/l
Percentage of time in the postoperative period with sensor glucose levels above target range | 1-2 weeks
  Proportion of time in the postoperative period with sensor glucose levels above 10.0mmol/l
Mean sensor glucose value in the preoperative period | 1 week
  Mean value of the sensor glucose levels in the preoperative period
Mean sensor glucose value in the perioperative period | 1 day
  Mean value of the sensor glucose levels in the perioperative period
Mean sensor glucose value in the postoperative period | 1-2 weeks
  Mean value of the sensor glucose levels in the postoperative period
Standard deviation of sensor glucose levels in the preoperative period | 1 week
  Standard Deviation of the sensor glucose levels in the preoperative period
Standard deviation of sensor glucose levels in the perioperative period | 1 day
  Standard Deviation of the sensor glucose levels in the perioperative period
Standard deviation of sensor glucose levels in the postoperative period | 1-2 weeks
  Standard Deviation of the sensor glucose levels in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD PhD, Principal Investigator — Inselspital, University Hospital of Bern, University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland